CLINICAL TRIAL: NCT05786885
Title: Microneedling With Vitamin C Versus Injectable Vitamin C for Depigmentation in Physiological Gingival Melanin Hyperpigmentation: A Randomized Controlled Clinical Trial
Brief Title: Microneedling With Vitamin C Versus Injectable Vitamin C for Depigmentation in Gingival Melanin Hyperpigmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Gamil, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22091990
Record Dates: First submitted 2023-03-05; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Gingival Pigmentation
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Microneedling will be done with application of topical vitamin C paste for depigmentation
  Interventions: Procedure: Microneedling will be done with application of topical vitamin C paste for depigmentation
- Control Group (Active Comparator): Gingival depigmentation will be done by vitamin C injection only.
  Interventions: Procedure: Vitamin C injection

INTERVENTIONS:
Procedure: Microneedling will be done with application of topical vitamin C paste for depigmentation — A Dermapen device will be used to microneedle the gingival tissue (model M8) with 24 microneedles arranged in rows, which is adjusted with 1.5 mm depth at the 6th mode speed of 700 cycles/min.
  It will be used in intermittent motion on the affected area for 30-40 seconds / tooth.
  Once bleeding points are observed on all areas of the pigmented gingiva, it will be irrigated using saline solution and dried using sterile gauze.
  Topical vitamin C powder (1000 mg/ml) will be mixed with saline, and the resultant slurry mix will then be applied to the gingiva for 10 minutes.
  Arms: Intervention Group
Procedure: Vitamin C injection — 1-1.5 ml Vitamin C will be injected into the gingiva, using an insulin syringe, once weekly, for 3 weeks.
  All the injection procedures will be performed by the same operator. The treated area will be left without dressing in both groups.
  Arms: Control Group

SUMMARY:
The study is a randomized controlled clinical trial comparing the use of microneedling with vitamin C against injecting vitamin C for depigmentation in physiological gingival melanin hyperpigmentation in a group of patients attending the outpatient clinic of the department of Oral Medicine and Periodontology-Cairo University.

DETAILED DESCRIPTION:
Melanin hyperpigmentation has been linked to a number of etiological and pathological causes, including smoking, heavy metal toxicity, heredity, endocrine disorders, UV exposure, inflammation, benign and malignant lesions, and intentional cultural tattooing. In order to determine whether the reason is physiological or pathological, a thorough medical history of the patient is essential.

With the introduction of gingival depigmentation as a periodontal surgical procedure, the hyperpigmented gingival tissues are removed utilizing a variety of surgical treatment methods, such as scalpel excision, bur abrasion, free gingival grafts, ADMA, lasers, cryosurgery, electro surgery.

The surgical approaches, albeit the most popular, are associated by anxiety, bleeding, a significant postoperative wound, and recurrence. Those methods could also have negative consequences include chemical burns, delayed healing, extreme pain and suffering, bone loss, and trouble controlling the depth of de-epithelization.

Vitamin C has been developed as a treatment for melanin pigmentation, due to its suppression of tyrosine activity, which directly downregulates dopaquinone synthesis, a precursor in the manufacture of melanin, as well as its epigenetic inhibitory effect on genes involved in melanocyte function. In vivo studies showed its impact on melanocyte function and quantitative productivity as well as how it affected melanocyte and keratinocyte cell-to-cell contact in a dose-dependent manner.

Local application of vitamin C to the gingiva as an adjunct to surgical depigmentation techniques has been shown in several case studies to depigment the gingiva or delay the repigmentation of the gingiva, supporting the possibility of using Vitamin C alone as a treatment modality for melanin-related gingival hyperpigmentation. In a study comparing the use of vitamin C injections versus the conventional surgical method, a statistical significant difference between both groups was found at one month regarding the mean values of changes in pigmentation index.

Needle-based delivery systems are designed to deliver medications by rupturing the skin or mucosal barrier, making the medication easily accessible to the targeted tissues. The collagen induction therapy method known as microneedling approach involves puncturing the skin repeatedly. Microneedling has been widely used in dermatology recently since it is a method that is efficient, straightforward, affordable, well-tolerated, and advantageous from both a cosmetic and therapeutic standpoint.

Instead of cutting through the cells, the used microneedles create microconduits that increase the skin's permeability and blood flow into the epidermis. This procedure makes it easier for topical drugs to cross the stratum corneum layer. Additionally, growth factors that support the regeneration of collagen and elastin are created.

The microneedling principle is suggested to be used in the treatment of gingival hyperpigmentation, compared to the currently employed techniques such as scalpel surgery, laser ablation, bur abrasion, and electrocautery which frequently result in complications, microneedling could be a promising minimally invasive, straightforward, painless, and cost-effective treatment modality for gingival depigmentation. Subsequent randomized controlled clinical trials are required to validate the findings for the case report that mentioned the use of Dermapen with vitamin C topical paste as a novel technique for gingival depigmentation.

Vitamin C has the ability to suppress tyrosine activity, which directly downregulates dopaquinone synthesis, a precursor in the manufacture of melanin, as well as its epigenetic inhibitory effect on genes involved in melanocyte function. Thus, Vitamin C injections can be used as a minimal invasive technique for physiological gingival melanin hyperpigmentation.

Microneedling has been widely used in dermatology due to its ability to create microconduits that increase the skin's permeability and blood flow into the epidermis. Thus, Dermapen together with vitamin C topical paste has been used as a novel technique for gingival depigmentation in a case report.

ELIGIBILITY:
Inclusion Criteria:

* Patients exhibiting physiological melanin hyperpigmentation in the anterior region of the upper or lower gingiva.
* Patients should be free from any systemic diseases according to modified Cornell Medical index.
* Non- smokers.

Exclusion Criteria:

* Patients with periodontal disease.
* Patients with endocrine disorders causing hyperpigmentation or drug induced gingival pigmentation.
* Pregnant or lactating females.
* Patients with known hypersensitivity to vitamin C.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Surface area of pigmentation | Measured at baseline
  an intraoral picture (labial view) showing the hyperpigmented gingiva of the patient, is uploaded to ImageJ software. the length of central incisor is measured intra orally from the incisal edge to the CEJ and used as a reference to adjust the image scale of the software. On ImageJ software, a line is drawn surrounding the pigmented area and the software automatically measures the surface area of the selected pigmented area
Surface area of pigmentation | Measured at 3 months after the intervention.
  an intraoral picture (labial view) showing the hyperpigmented gingiva of the patient, is uploaded to ImageJ software. the length of central incisor is measured intra orally from the incisal edge to the CEJ and used as a reference to adjust the image scale of the software. On ImageJ software, a line is drawn surrounding the pigmented area and the software automatically measures the surface area of the selected pigmented area

SECONDARY OUTCOMES:
Dummett-Gupta Oral Pigmentation Index | Measured at baseline and 3 months after the intervention.
  The degree of gingival pigmentation is scored as 0, pink tissue [no clinical pigmentation]; 1 = mild light brown tissue [mild clinical pigmentation]; 2, medium brown or mixed brown and pink tissue [moderate clinical pigmentation]; or 3, deep brown/blue-black tissue [heavy clinical pigmentation].
Gingival thickness | Measured at baseline and 3 months after the intervention.
  Using a standard no. 35 endodontic finger spreader with a rubber stop. The gingival biotype will be considered thin if the measurement is ≤1.0 mm and thick if it measured >1.0 mm.
Pain (patient related outcome) | Recorded daily, starting from the same day after the intervention, up to 7 days after the intervention.
  Using Visual analogue score questionnaire, score is from 0-10, where 0 is the minimum value representing no pain and 10 is the maximum value representing the highest level of pain felt.
Pain (patient related outcome) | 7 days after the intervention.
  The rate of analgesic consumption will be recorded.
Patient Satisfaction | Measured 3 months after the intervention.
  Using questionnaire to score the degree of patient satisfaction with the cosmetic results of the procedure. It will be documented depending on the patient's opinion, measured on a five-point scale 0: Very dissatisfied 1: Dissatisfied 2: Neither satisfied nor dissatisfied 3: Satisfied 4: Very satisfied